CLINICAL TRIAL: NCT00237146
Title: Study to Evaluate Zoledronic Acid on Quality of Life and Skeletal-related Events as Adjuvant Treatment in Patients With Hormone-naïve Prostate Cancer and Bone Metastasis Who Have Undergone Orchiectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EVE01
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Zoledronic acid; Bone metastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- Zoledronic Acid (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
An open, multicenter and prospective study to evaluate the impact of the treatment with zoledronic acid 4 mg, on the quality of life and the skeletal-related events in patients with prostate cancer and bone metastasis that responds to hormonal therapy. Zoledronic acid is given to patients in a 15 minute-infusion every 4 weeks until a skeletal-related event occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* histologically confirmed adenocarcinoma of the prostate.
* Orchidectomy within the four previous weeks to enter the study.
* bone metastasis evidenced by bone scan.
* A hip DEXA study with a DS < 3.
* No hormonal therapy previous to enter the study.
* ECOG performance score of 0-2.
* Signed written informed consent.

Exclusion Criteria:

* Abnormal renal function evidenced by a creatinine clearance ≤60 ml/min.
* Any kind of hormonal therapy for prostate cancer previous to enter the study.
* Serum calcium corrected for albumin level < 8.0 mg/dl.
* WBC < 3.0x10^3, ANC < 1500/mm3, Hemoglobin < 8.0 g/dl, platelets < 75 x 10^3/l.
* Abnormal hepatic function evidenced by ALT and AST value >2.5 UNL
* Subjects with any other malignant disease that can affect the bone.
* Subjects with any other non malignant disease that can jeopardize the evaluation of the primary objectives of this trial (severe osteoporosis) or that do not aloud perform the trial evaluations.
* Known hypersensibility to zoledronic acid or other bisphosphonates.
* Subjects that in the investigator's opinion can not cooperate with the protocol.

Other protocol inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of Zometa® (Zoledronic Acid) i.v in doses of 4mg for measure the following parameters of efficacy: Quality of Life, Incidence of Events related to the skeleton

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Caracas, Venezuela